CLINICAL TRIAL: NCT06348056
Title: A Comparison of the Metabolic Effects of Zinc-Amino Acid (ZnAA) Versus Zinc Gluconate Given in a Fasted State
Brief Title: A Comparison of the Metabolic Effects of Zinc-Amino Acid (ZnAA) Versus Zinc Gluconate
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2022-07-15499
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Response of Fatty Acid Desaturation to Zinc Intake

STUDY DESIGN:
Intervention Model Description: Participants will take the first zinc supplement for two weeks, followed by a two-week washout period, and then take the second zinc supplement for two weeks. The order of whether the first supplement is the zinc amino acid complex, or zinc gluconate, will be randomized.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The two zinc supplements will have the same appearance, and will be in coded bottles, such that the participant, care provider, investigator, and outcomes assessor may be kept unaware of the order of the supplements for each participant until the data analysis is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zinc Amino Acid (Experimental): The zinc in the supplement is complexed with the amino acids lysine and glutamate.
  Interventions: Dietary Supplement: 30 mg Zn Amino Acid daily for 13 days
- Zinc Gluconate (Experimental): The zinc in the supplement is complexed with gluconate.
  Interventions: Dietary Supplement: 30 mg Zn Gluconate daily for 13 days

INTERVENTIONS:
Dietary Supplement: 30 mg Zn Amino Acid daily for 13 days — A 30 mg zinc amino acid supplement is taken p.o. in the fasted state for 13 days.
  Arms: Zinc Amino Acid
Dietary Supplement: 30 mg Zn Gluconate daily for 13 days — A 30 mg zinc gluconate supplement is taken p.o. in the fasted state for 13 days.
  Arms: Zinc Gluconate

SUMMARY:
Food consumption affects zinc metabolism within the body. Lowe and colleagues demonstrated that zinc is directed out of plasma and into tissues, such as into the liver, postprandially . It is likely that zinc absorbed with a meal is directed to the liver via the portal circulation whereas that zinc taken in the fasted state is more readily directed to peripheral blood plasma. Zinc taken with food is more likely to be bound to components of the food matrix and, therefore, it is not absorbed as efficiently by Zip4 ionic zinc transporters in the upper gastrointestinal tract. Some of the zinc in the food matrix may, however, be co-absorbed with amino acids over the whole length of the small intestine . Co-absorption of zinc with amino acids may explain the greater effects of zinc taken with food on omega-6 fatty acid desaturation . The investigators propose that this effect may be maximized by providing supplemental zinc complexed with amino acids. Since the zinc amino acid complex likely mimics the absorption and retention of zinc bound to protein in food, the investigators further propose that zinc, bound to amino acids taken in the fasted state will be directed into the cellular compartments more efficiently than zinc associated with gluconate.

The primary aim in this study is to determine whether providing a zinc amino acid complex has a greater effect on indices of essential fatty acid desaturation compared with zinc gluconate when the zinc complexes are taken in the fasting state.

The investigators hypothesize that taking a zinc amino acid (Zn-AA) complex in a fasted state daily for two weeks has a greater effect on the Fatty Acid Desaturase 1 (FADS1) activity compared with zinc gluconate. Also, if the uptake of ionic zinc gluconate into cellular compartments is reduced in comparison to Zn-AA because the zinc gluconate is retained in the plasma, two weeks of a daily zinc gluconate will have a greater effect on fasting plasma zinc concentrations compared to a Zn- AA complex.

DETAILED DESCRIPTION:
Once the informed consent is obtained and the schedule is set with the participant, the participant will pick up their zinc bottle they will consume for the first two weeks and will start the study on the scheduled date.

Visit 1 (Week 1, Day 1): The participants will come to Morgan Hall fasting for their first blood draw visit. They will come to the clinic after an 8-hour fast and we will collect a blood sample. They will be instructed to take their zinc starting on day 2 every morning thirty minutes prior to having their regular breakfast and to write what they eat for breakfast in their breakfast log daily. They will take the given zinc for thirteen days (days 2-14).

Visit 2 (Week 2, Day 15): The participants will come to Morgan Hall after an 8-hour fast and the investigators will collect a second blood sample. Subjects will then be given instructions for visits three and four which will take place two weeks later to allow for a washout period between the crossover studies.

Visit 3 (Week 5, Day 1): The participants will come to Morgan Hall fasting for their third blood draw visit. They will come to the clinic after an 8-hour fast and the investigators will collect a blood sample. Subjects will be instructed to take the alternate zinc starting on day 2 every morning thirty minutes prior to having their regular breakfast and to record their breakfast in their breakfast log daily. They will take the given zinc for thirteen days (days 2-14).

Visit 4: (Week 6, Day 15): The participants will come to Morgan Hall after an 8-hour fast and the investigators will collect a final fourth blood sample. The subjects' breakfast logs will be collected at this time and their participation in the study will be completed.

Study diets:

Study subjects will receive a total of 26 days of zinc (13 days of one form prior to the washout period, and then 13 of the alternate form after). They will be provided with 13 days of zinc 30 mg zinc, as zinc gluconate, and 30 mg zinc, as a zinc amino acid complex, per day. They will be randomly assigned to which form of zinc they will take for the first two weeks, taking either zinc gluconate or zinc amino acid in a fasted state. All participants will be asked to take the zinc in the fasted state at least 30 minutes before their breakfast meal. The men will log their breakfast foods, the amounts consumed, and the time they ate breakfast every day. They will be asked to maintain a steady dietary pattern over the course of the two weeks as well as maintain a steady physical activity routine.

Fasting:

No food is allowed for an 8-hour period before any of the 4 visits requiring blood sampling. Water can and should be consumed during the fast to maintain hydration and to facilitate blood collection. Any other beverages besides water are not to be consumed during the fasting period.

Blood samples (week 1, day 1; week 2, day 15; week 5, day 1; week 6, day 15.) Participants will provide a total of 4 blood samples during the study. The blood sample will be drawn by inserting a needle into a vein in their arm. Each sample will be approximately 15 ml (or 1 tablespoon); a total of 60 ml (about 1/4 cup) will be drawn for the whole study.

Laboratory analysis of samples. Blood samples will be analyzed for their total zinc content by inductively coupled plasma - optical emission spectrometry (ICP-OES) and for FADS1 activity index along with other fatty acids by liquid chromatography with tandem mass spectrometry (LC-MS/MS).

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy men (i.e., have no current health issues requiring medications or a specific diet)
* 18 to 50 years of age
* Body mass index between 18 and 30 kg/m2
* Willing to take zinc supplements provided by the study for a total of four weeks

Exclusion Criteria:

* History of heart disease, any inflammatory disorder including inflammatory bowel syndrome or arthritis, or any cancer treatment, or previously diagnosed with HIV
* Smoking or alcohol abuse, use of illicit drugs
* Any contraindication to venipuncture such as bleeding disorders or use of blood thinners
* Those taking vitamins or supplements including minerals and omega oils, who cannot agree to stop taking the supplements two weeks prior to the study and for the duration of the study

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
FADS1 activity index | Day 1 (baseline 1), day 15 (endpoint 1), day 29 (baseline 2), day 43 (endpoint 2)
  The molar ratio (unitless) of arachidonic acid to dihomo-gamma-linolenic acid, i.e., fatty acid desaturase 1 (FADS1) product to precursor.

SECONDARY OUTCOMES:
Fasted plasma zinc concentration | Day 1 (baseline 1), day 15 (endpoint 1), day 29 (baseline 2), day 43 (endpoint 2)
  The concentration of zinc in blood plasma (mg/dL) sampled following an overnight fast

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Berkeley, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data on FADS1 activity index and plasma zinc concentration will be made available upon request.